CLINICAL TRIAL: NCT01573884
Title: Ex Vivo Exploratory Analysis in Healthy Full-term Infants
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: AK97
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Last update posted 2012-04-10 (Estimated); Status verified 2012-04

CONDITIONS: Healthy Infant and Mother Pairs

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
* Exploratory analyses of the immune response in a ex vivo culture system
* Characterization of the composition of maternal milk and infant urine

ELIGIBILITY:
Inclusion Criteria

* Infant or infant-mother pair in good health
* Infant or infant-mother pair is from smoke-free home
* Infant is a singleton, full term
* birth weight was > 2490 g
* Between 0 and 17 days of age at enrollment
* Human milk fed infants must have been exclusively human milk-fed since birth; formula fed infants must have received Similac Advance or Similac Sensitive since birth
* Parents confirm their intention not to administer vitamin or mineral supplements (excluding vitamin or mineral supplements containing vitamin D), solid foods or juices to their infant from enrollment throughout the study

Exclusion Criteria:

* An adverse maternal, fetal or infant medical history, including gestational diabetes that is thought by the investigator to have potential for effects on tolerance, growth, and/or development.
* Infant has been treated with antibiotics
* Participation in another study -

Max Age: 17 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: infant and mother pairs
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Viral load in cell cultures | 14 days

SECONDARY OUTCOMES:
Changes in viral load and cytokine profiles | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Karen Goehring, MS, Study Chair — Abbott Nutrition
Locations (2):
- United States (2):
  - Northpoint Pediatrics, Indianapolis, Indiana
  - Institute of Clinical Research, Mayfield Heights, Ohio